CLINICAL TRIAL: NCT04407819
Title: Sarcopenia and Diabetes Mellitus
Acronym: SARCoDM
Status: Completed | Type: Observational
Sponsor: Dionyssiotis, Yannis, M.D. (Individual)
Collaborators: University of Thessaly (Other)
Responsible Party: Principal Investigator, Yannis Dionyssiotis, Post graduate student in Hellenic Open University of Greece, Dionyssiotis, Yannis, M.D.
Other Study IDs: EAPDionyssiotis
Record Dates: First submitted 2020-05-19; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Sarcopenia
Keywords: sarcopenia; diabetes mellitus; skeletal muscle index
MeSH Terms: conditions — Sarcopenia; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetes mellitus type 2: 36 patients with diabetes mellitus type 2, aged 20-80 years, attending endocrinology outpatient clinics were studied for the assessment of muscle mass and function compared to controls.
  Interventions: Radiation: WHOLE BODY DXA
- CONTROLS: 14 community people who visited the endocrinology outpatient hospital clinic for a routine checkup, or with a non-related to diabetes disease.
  Interventions: Radiation: WHOLE BODY DXA

INTERVENTIONS:
Radiation: WHOLE BODY DXA — Muscle mass was estimated by using the whole body DXA (Hologic Horizon W)

SUMMARY:
The association of diabetes mellitus type 2 (T2DM) with sarcopenia has not been adequately investigated. Sarcopenia is characterized by progressive and generalized loss of skeletal muscle mass which may affect performance.

DETAILED DESCRIPTION:
The relationship between DM and sarcopenia has not been extensively investigated. Skeletal muscle is the primary site of glucose deposition, and decreased muscle mass plays a role in impaired glucose metabolism in patients with insulin resistance and type 2 diabetes. Skeletal muscle resistance to insulin action appears to be the link between type 2 diabetes (T2DM) and sarcopenia. Hyperglycemia is a metabolic dysfunction which can potentially damage muscle cells. Insulin deficiency leads to marked muscle catabolism that can be reversed by exogenous insulin administration.

The metabolic disorder in diabetics may be reversible.Thus, it may be possible to restore physical ability by restoring the musculoskeletal system.Therefore, the diagnosis of sarcopenia if made can lead to interventions which may prevent the deterioration of body composition and the subsequent deterioration of quality of life. According to the results of the aforementioned studies it is still inconclusive if the metabolic disorder in diabetes may be related to sarcopenia, or sarcopenia may be a consequence of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* T2DM participants were on treatment with oral hypoglycemic agents
* confirmation criteria of a T2DM diagnosis were glycosylated hemoglobin A1c levels ≥ 6.5% and fasting plasma glucose ≥ 126 mg/dl (7 mmol/l).

Exclusion Criteria:

* history of a cerebrovascular event, a heart stent, an artificial cardiac pacemaker or other metallic implant,
* a malignant tumor, liver disease, end stage chronic kidney disease, a thyroid disorder, carpal tunnel syndrome,
* subjects who received special dietary supplements such as protein powder, during the last three months were excluded from the study.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A group of 36 patients, aged 20-80 years old, 18 male and 17 female with type 2 diabetes mellitus, and a control group with the same demographic characteristics, participated in the study. All were previously examined by an endocrinologist (in a public hospital, private or university outpatient clinic) from March to July 2018. The control group consisted of 14 community people who visited the endocrinology outpatient hospital clinic for a routine checkup, or with a non-related to diabetes disease.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-09-22 (Actual)

PRIMARY OUTCOMES:
Skeletal Muscle Index | Up to 12 weeks
  Appendicular Muscle Mass/Height2
prevalence of sarcopenia in patients with T2D and in the control group | Up to 12 weeks
  percents in different groups

SECONDARY OUTCOMES:
fat mass | Up to 12 weeks
  percent of fat mass, Total Fat index

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Dionyssiotis, MD, PhD, Principal Investigator — Foundation for Care of Neurological Illnesses, Greece
Locations (1):
- Foundation for Care of Neurological Illnesses, Greece, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dionyssiotis Y. Sarcopenia in the Elderly. Eur Endocrinol. 2019 Apr;15(1):13-14. doi: 10.17925/EE.2019.15.1.13. Epub 2019 Apr 12. PMID 31244904
- [Background] Dionyssiotis Y, Kapsokoulou A, Samlidi E, Angoules AG, Papathanasiou J, Chronopoulos E, Kostoglou-Athanassiou I, Trovas G. Sarcopenia: From definition to treatment. Hormones (Athens). 2017 Oct;16(4):429-439. doi: 10.14310/horm.2002.1764. No abstract available. PMID 29518764